CLINICAL TRIAL: NCT01370694
Title: An Open-Label, Single Arm Study of MK-8808 in Patients With Advanced CD20-Positive Follicular Lymphoma
Brief Title: Study of MK-8808 for Participants With Follicular Lymphoma (MK-8808-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated for business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8808-001; 2011-000386-13 (EudraCT Number)
Record Dates: First submitted 2011-05-18; First posted 2011-06-10 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Cyclophosphamide; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-8808 Combination Therapy (Experimental): Participants received MK-8808 375 mg/m^2 intravenously (IV) + cyclophosphamide 750 mg/m^2 IV + vincristine 1.4 mg/m^2 IV (maximum dose of 2 mg IV) on Day 1 each cycle, plus prednisolone 40 mg/m^2, orally on Days 1 to 5 of each cycle for a maximum of 8 cycles. Participants receiving clinical benefit could remain on MK-8808 375 mg/m^2 IV starting 8 weeks after last dose of combination therapy, every 2 months for up to 2 years.
  Interventions: Drug: MK-8808; Drug: cyclophosphamide; Drug: vincristine; Drug: prednisolone

INTERVENTIONS:
Drug: MK-8808
Drug: cyclophosphamide
Drug: vincristine
Drug: prednisolone

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and anti-tumor activity of MK-8808 in combination with cyclophosphamide, vincristine, and prednisolone (CVP), and as a single agent, for participants with B-lymphocyte antigen cluster of differentiation 20 (CD20)-positive follicular lymphoma who have had no prior chemotherapy. The primary study hypothesis is that MK-8808 will be safe and well tolerated in combination with CVP and as a single agent.

DETAILED DESCRIPTION:
The study was terminated early by the Sponsor due to business reasons. All participants were discontinued from MK-8808 + CVP, but could continue to receive maintenance therapy with MabThera™ (rituximab) per standard of care.

ELIGIBILITY:
Inclusion criteria:

* Histological diagnosis of CD20-positive follicular lymphoma, Grade 1, 2, or 3a (World Health Organization [WHO] 2008 classification) based on an excisional or incisional lymph node biopsy or a bone marrow biopsy.
* Ann Arbor Stage III or IV disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Life expectancy >3 months with no expected need of immediate intervention to treat life-threatening complications.
* Adequate organ function.
* Participants must agree to use an adequate method of contraception starting with the first dose of study drug through 12 months (for females) or 90 days (for males) after the last dose of study drug.

Exclusion criteria:

* Histological Grade 3b or with >50% diffuse architectural pattern.
* Circulating malignant cells >25,000/mm^3
* Presence or history of central nervous system (CNS) disease (either CNS lymphoma or lymphomatous meningitis).
* Prior treatment with chemotherapy, rituximab, any other anti-CD20 compound, or any other type of anti-cancer compounds.
* Radiotherapy within 2 months prior to Cycle 1 Day 1.
* Current participation or has participated in a study with an investigational compound within 30 days prior to Cycle 1 Day 1.
* Concomitant disease that requires continuous therapy with prednisone at doses >20 mg per day.
* Any medical contraindication for prednisolone as being dosed in the CVP regimen.
* Poorly controlled diabetes mellitus, as defined by institutional or local standards.
* Grade >2 peripheral neuropathy.
* Has one of the following:

  1. is human immunodeficiency virus (HIV)-positive
  2. is Hepatitis B surface antigen positive (HBsAg+) or is positive for antibodies to Hepatitis B core antigen (anti-HBcAg+)
  3. has antibodies to Hepatitis C virus
* Has one or more of the following:

  1. Active tuberculosis based on institutional diagnostic criteria and local practice guidelines.
  2. Evidence of a tuberculosis infection based on a chest X-ray (CXR) or computed tomography (CT) scan performed within 3 months of dosing.
  3. History of a tuberculosis infection.
* Major surgical procedure within 4 weeks prior to Cycle 1 Day 1.
* Regular use (including "recreational" use) of any illicit drugs or recent history (within the last year) of drug or alcohol abuse or dependence.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-08-19 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/study.html?id=8808-001&kw=8808-001&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated early by the Sponsor due to business reasons. All participants were discontinued from MK-8808 on 18 March 2014, but could continue to receive maintenance therapy with rituximab per standard of care.
Period: Overall Study
Arm/Group | MK-8808 Combination Therapy
Started | 7
Completed | 1
Not Completed | 6
Not completed — Switched to rituximab | 4
Not completed — Progressive disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | MK-8808 Combination Therapy
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Clinical and Laboratory Adverse Events (AEs) During MK-8808/CVP Combination Therapy
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment.
Time Frame: From first dose of combination therapy up to 24 weeks
Population: All participants receiving at least one dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | MK-8808 Combination Therapy
Number analyzed (Participants) | 7
Participants | 6

2. Primary Outcome: Number of Participants Experiencing Clinical and Laboratory AEs During MK-8808 Maintenance Therapy
Description: as for outcome 1
Time Frame: From first dose of single agent MK-8808 up to 2 years
Population: No participants progressed to MK-8808 single agent maintenance therapy; this outcome measure was not assessed.
Arm/Group | MK-8808 Combination Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Maximum Concentration (Cmax) of Plasma Levels of MK-8808 When Used in Combination With CVP
Description: Cmax is a measure of the maximum concentration of the drug in the plasma as measured using plasma samples taken over specified time points.
Time Frame: Pre-dose and end of infusion in each 21-day cycle and at end of therapy visit (up to 24 weeks)
Population: This analysis was not done due to early termination of the study.
Arm/Group | MK-8808 Combination Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Cmax of Plasma Levels of MK-8808 During Single Agent Maintenance Therapy
Description: Cmax is a measure of the maximum amount of drug in the plasma over time using samples taken at specified time points.
Time Frame: Predose and end of infusion in every other cycle and at end of therapy visit (up to 2 years)
Population: No participants progressed to MK-8808 single agent maintenance therapy; this outcome measure was not assessed.
Arm/Group | MK-8808 Combination Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Lowest Concentration (Ctrough) of Plasma Levels of MK-8808 When Used in Combination With CVP
Description: Ctrough is a measure of the lowest level of drug in the plasma over time, using plasma samples collected at specified time points.
Time Frame: Pre-dose and end of infusion in each 21-day cycle and at end of therapy visit (up to 24 weeks)
Population: This analysis was not done due to early termination of the study.
Arm/Group | MK-8808 Combination Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Ctrough of Plasma Levels of MK-8808 When Used as Single Agent Maintenance
Description: as for outcome 5
Time Frame: Predose and end of infusion in every other cycle and at end of therapy visit (up to 2 years)
Population: No participants progressed to MK-8808 single agent maintenance therapy; this outcome measure was not assessed.
Arm/Group | MK-8808 Combination Therapy
Number analyzed (Participants) | 0

7. Secondary Outcome: Clinical Response of Tumor to MK-8808/CVP Combination Therapy
Description: The response of the tumor to MK-8808/CVP combination therapy was radiographically assessed using Response Criteria Evaluation in Solid Tumors (RECIST). Response categories of partial response (PR), complete resonse (CR), and uncomfirmed (CRu) central review.
Time Frame: Up to 2 years
Population: All participants with evaluable data
Measure: Number; unit: Participants
Arm/Group | MK-8808 Combination Therapy
Number analyzed (Participants) | 7
Participants
  PR | 6
  CR | 0
  CRu | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of CVP therapy (up to 28 weeks)
Description: Adverse events were not collected for participants who were switched to MabThera.
Arm/Group | MK-8808 Combination Therapy
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8808 Combination Therapy (N=7)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8808 Combination Therapy (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated for business reasons. Not all planned analyses were performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.